CLINICAL TRIAL: NCT01446029
Title: Telemonitoring to Improve Outcomes of Patients With Chronic Kidney Disease
Brief Title: Telemonitoring to Improve Outcomes of Patients With Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Areef Ishani, Chief, Section of Nephrology; Associate Professor of Medicine, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Minn-VAMC-4292-A
Record Dates: First submitted 2011-09-28; First posted 2011-10-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Kidney Disease
Keywords: Telemonitoring; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention)
- Intervention Device (Active Comparator)
  Interventions: Device: Video Telemonitoring Device with Clinical Care Modules

INTERVENTIONS:
Device: Video Telemonitoring Device with Clinical Care Modules — Telemonitoring of vital signs; videoconferencing, remote titration of diabetes, blood pressure, and lipid medications using evidence based treatment algorithm, and cooperative goal setting using education modules to enhance lifestyle changes
  Other Names: Telehealth; Telemonitoring; Chronic Disease Management
  Arms: Intervention Device

SUMMARY:
The purpose of this study is to determine if the adoption of a chronic care model in conjunction with tele monitoring and case management can reduce the risk of death, hospitalization, emergency room visits, or admission to a skilled nursing facility in patients with chronic kidney disease compared to usual care.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major public health issue. Approximately, 11% of the US population has CKD with an increased prevalence among individuals great than 65years. Many individuals with CKD go unrecognized because they are typically asymptomatic. Individuals with CKD have been demonstrated to have a greater risk for mortality, hospitalization and development of end stage kidney disease. Also, individuals with CKD consume a significantly greater proportion of health care expenditures compared to other patients. This study aims to determine if the adoption of a chronic care model in conjunction with telemonitoring and case management can reduce risk of death, hospitalization, ER visits or admission to a skilled nursing facility in patients with CKD compared to usual care. This study will use a randomized controlled trial. Few interventions have been demonstrated to improve clinical outcomes in patients with CKD. If successful, this study will enable the VA to provide high quality care to patients with CKD while potentially reducing the cost of providing care.

ELIGIBILITY:
Inclusion Criteria: Enrolled at Minneapolis or St. Cloud Veterans Affairs Health Care System (VAHCS) or affiliated Community Based Outcomes Clinic(CBOC); Late eGFR within the VA system <60 ml/min/1.73m2 -

Exclusion Criteria: Primary care provider unwilling to have participant included in study; unable to give consent; severe mental health condition; living in a nursing home

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
composite clinical outcome (reduce risk of death, hospitalization, emergency room visits, admission to skilled nursing facility) | one year

SECONDARY OUTCOMES:
reduction of cost | one year
incidence of end stage kidney disease | one year
hospital re-admission | one year
Intervention group achieving National Kidney guideline values for blood pressure, glycemia, lipids, and hemoglobin | one year

CONTACTS AND LOCATIONS:
Overall Officials: Areef Ishani, MD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- VA Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Barrett BJ, Garg AX, Goeree R, Levin A, Molzahn A, Rigatto C, Singer J, Soltys G, Soroka S, Ayers D, Parfrey PS. A nurse-coordinated model of care versus usual care for stage 3/4 chronic kidney disease in the community: a randomized controlled trial. Clin J Am Soc Nephrol. 2011 Jun;6(6):1241-7. doi: 10.2215/CJN.07160810. Epub 2011 May 26. PMID 21617090
- [Background] Ishani A, Greer N, Taylor BC, Kubes L, Cole P, Atwood M, Clothier B, Ercan-Fang N. Effect of nurse case management compared with usual care on controlling cardiovascular risk factors in patients with diabetes: a randomized controlled trial. Diabetes Care. 2011 Aug;34(8):1689-94. doi: 10.2337/dc10-2121. Epub 2011 Jun 2. PMID 21636796
- [Background] Santschi V, Chiolero A, Burnand B, Colosimo AL, Paradis G. Impact of pharmacist care in the management of cardiovascular disease risk factors: a systematic review and meta-analysis of randomized trials. Arch Intern Med. 2011 Sep 12;171(16):1441-53. doi: 10.1001/archinternmed.2011.399. PMID 21911628